CLINICAL TRIAL: NCT01008007
Title: Effect of VIUSID Administration on Adults With Acute Fever of Viral Etiology
Brief Title: Viusid in Adults With Acute Fever of Viral Etiology
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Mayra R. Carrasco García, "Salvador Allende" Clinical-Surgical Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAT-0911-CU
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Acute Fever of Viral Etiology
Keywords: Viusid; Dietary supplements; Acute fever; Viral etiology
MeSH Terms: interventions — Viusid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Viusid in combination with the conventional treatment for acute fever of viral etiology
  Interventions: Dietary Supplement: Viusid
- B (Active Comparator): Conventional treatment for acute fever of viral etiology
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Dietary Supplement: Viusid — One Viusid bag (4 grams, orally administered) every 8 hours, for 6 days in combination with the conventional treatment consisting in: intramuscular injection of one bulb of Dipyrone (600 mg) every 8 hours if fever is greater or equal to 38 ºC; intramuscular injection of one bulb of dimenhydrinate (50 mg) every 8 hours if vomiting; oral rehydration solution (8 ounce) after each diarrhea.
  Arms: A
Drug: Conventional treatment — Conventional treatment consisting in: intramuscular injection of one bulb of Dipyrone (600 mg) every 8 hours if fever is greater or equal to 38 ºC; intramuscular injection of one bulb of dimenhydrinate (50 mg) every 8 hours if vomiting; oral rehydration solution (8 ounce) after each diarrhea.
  Arms: B

SUMMARY:
The purpose of the study is to assess the safety and effect of Viusid (bags of 4 grams) administration in the treatment of acute fever of viral etiology as diagnosed by clinical, hematologic and serologic parameters. The duration of this open and randomized phase 2 clinical trial will be 6 days. The estimated number of persons with acute fever of viral etiology to be recruited and randomized for the study is 200. The primary outcome measure: platelet, leukocyte and granulocyte count will be assessed at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Acute fever of viral etiology with less than 72 hours of progression
* Signed informed consent.

Exclusion Criteria:

* Patients under treatment with other antioxidants.
* Inability to swallow the content of Viusid bags

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The platelet count improvement at 6 days (end of the treatment) | 6 days
The leukocyte count improvement at 6 days (end of the treatment) | 6 days
The granulocyte count improvement at 6 days (end of the treatment) | 6 days

SECONDARY OUTCOMES:
Clinical symptoms disappear during the Viusid administration (6 days). | 6 days
Adverse effects during treatment | 6 days
Hemoglobin level improvement | 6 days
Hematocrit level improvement at 6 days (end of the treatment) | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Mayra R Carrasco García, MD, Principal Investigator — "Salvador Allende" Clinical-Surgical Hospital
Locations (1):
- "Salvador Allende" Clinical-Surgical Hospital, Havana, La Habana, Cuba